CLINICAL TRIAL: NCT01085279
Title: Non-ablative 1,550 nm Fractional Laser Therapy Versus Triple Topical Therapy for the Treatment of Melasma: a Randomized Controlled Split-face Study
Brief Title: Fractional Laser as Treatment Option for Various Pigment Disorders (Fractional-3)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Responsible Party: Albert Wolkerstorfer, MD PhD, Netherlands Institute for Pigment Disorders
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fractional-3
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Pigmentation Disorder
Keywords: fractional laser; melasma; topical bleaching
MeSH Terms: conditions — Pigmentation Disorders; Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-ablative fractional laser (Experimental): In each patient, one side of the face was treated with non-ablative fractional laser in four-five sessions.
  Note: this study had a split-face design. In each patient, each side of the face was randomized to receive either non-ablative fractional laser therapy or triple topical therapy.
  Interventions: Device: Fraxel Restore, Solta Medical Inc. (Non-ablative fractional laser)
- Triple topical therapy (Active Comparator): In each patient, one side of the face was treated with triple topical therapy (Hydroquinone 5%, tretinoin 0.05%, triamcinolone acetonide 0.1%) during 15 weeks.
  Note: this study had a split-face design. In each patient, each side of the face was randomized to receive either non-ablative fractional laser therapy or triple topical therapy.
  Interventions: Drug: Modified Kligman's formula (Triple topical therapy)

INTERVENTIONS:
Device: Fraxel Restore, Solta Medical Inc. (Non-ablative fractional laser) — 1,550 nm non-ablative fractional laser Irradiance: 15 mJ/microbeam. Coverage: 14-20%. Number of treatment sessions: 4-5
  Other Names: Fraxel re:store, Solta Medical Inc., Hayward, CA
  Arms: Non-ablative fractional laser
Drug: Modified Kligman's formula (Triple topical therapy) — Hydroquinone 5%, tretinoin 0.05%, triamcinolone acetonide 0.1% once a day during 15 weeks
  Other Names: modified Kligman formula
  Arms: Triple topical therapy

SUMMARY:
The purpose of this study is to determine whether the use of non-ablative fractional laser is safe and effective in the treatment of melasma.

ELIGIBILITY:
Inclusion Criteria:

* Melasma
* Subjects attending the outpatient department of the Netherlands Institute for Pigment Disorders
* Age at least 18 years
* Subject is willing and able to give written informed consent

Exclusion Criteria:

* use of bleaching creams during the past six weeks
* history of keloid
* active eczema
* suspected hypersensitivity to lidocaine or triple therapy
* use of isotretinoin in the past six months
* high exposure of the lesion to sunlight or UV light (UVA or UVB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Physician's global assessment | T0, 3 weeks, and 3 and 6 months follow-up
  Improvement of hyperpigmentation was assessed by an independent blinded dermatologist. The results were scored on a scale from zero to six (0: total clearance (100% improvement), 1: almost total clearance (90-99% improvement), 2: distinct clearance (75-89% improvement) 3: moderate clearance (50-74% improvement) 4: mild clearance (25-49% improvement) 5: no change, 6: worsening of hyperpigmentation).

SECONDARY OUTCOMES:
L-value | T0, 3 weeks and 3 and 6 months follow-up
  Improvement of hyperpigmentation was assessed by color measurement through reflectance spectroscopy (Microflash 200 d, Datacolor International, Lawrenceville, GA). This instrument, with an aperture of 4 mm, determines color by measuring the intensity of reflected light of particular wavelengths. In this study, the obtained L value, indicating the lightness of the measured area of skin, was used.
Melanin index | T0, 3 weeks and 3, and 6 months follow-up
  Melanin index was measured using a spectrometer (Derma-Spectrometer, Cortex Technology ApS, Hadsund, Denmark) in order to assess changes in the amount of dermal and epidermal melanin.
Patient's global assessment | 3 weeks, 3 and 6 months follow-up
  Patients were asked to score the improvement of hyperpigmentation on a visual analogue scale (VAS) from 0 to 10 (Patient's Global Assessment, PGA) at all follow-up moments.
Patient's satisfaction | 3 weeks, 3 and 6 months follow-up
  Patient's satisfaction was scored on a visual analogue scale (VAS) from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Wolkerstorfer, MD PhD, Principal Investigator — Netherlands Institute for Pigment Disorders
Locations (1):
- Netherlands Institute for Pigment disorders, Amsterdam, Netherlands